CLINICAL TRIAL: NCT02335489
Title: A Post Market Cohort to Assess the Performance of the Spinal Modulation Neurostimulator System for the Management of Chronic Neuropathic Pain of the Foot and/or Lower Leg
Status: Terminated | Type: Observational
Why Stopped: A significant local issue has to led to the suspension of recruitment, this study will be terminated in the coming months
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-SMI-2013
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Chronic Neuropathic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treated Subjects: All subjects recruited and treated with the Axium neurostimulator
  Interventions: Device: Implantation with the commercially available Axium neurostimulator

INTERVENTIONS:
Device: Implantation with the commercially available Axium neurostimulator

SUMMARY:
14-SMI-2013 is a post market, observational, questionnaire based study to assess the effectiveness of the commercially available Axium neurostimulator in the management of neuropathic pain of the foot and/or lower limb

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years old
2. Subject is able and willing to comply with the follow-up schedule and protocol
3. Chronic, intractable pain in the foot and/or lower leg for at least 6 months
4. Failed conservative treatments for chronic pain including but not limited to pharmacological therapy, physical therapy and interventional pain procedures for chronic pain
5. Minimum baseline pain rating of 60 mm on the Visual Analog Scale in the primary region of pain
6. Subject is able to provide written informed consent

Exclusion Criteria:

1. Female subject of childbearing potential is pregnant/nursing, plans to become pregnant or is unwilling to use approved birth control
2. Escalating or changing pain condition within the past month as evidenced by investigator examination
3. Subject has had corticosteroid therapy at an intended site of stimulation within the past 30 days
4. Subject has had radiofrequency treatment of an intended target Dorsal Root Ganglion within the past 3 months
5. Subject currently has an active implantable device including implantable cardioverter defibrillator, pacemaker, spinal cord stimulator or intrathecal drug pump
6. Subject is unable to operate the device
7. Subjects with indwelling devices that may pose an increased risk of infection
8. Subjects currently has an active infection
9. Subject has participated in another clinical investigation within 30 days
10. Subject has a coagulation disorder or uses anticoagulants that, in the opinion of the investigator, precludes participation
11. Subject has been diagnosed with cancer in the past 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Neuropathic Pain of the Foot and/or Lower Leg
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- AZ Nikolaas, Sint-Niklaas, Belgium

RESULTS

PARTICIPANT FLOW:
Groups:
- All Enrolled Subjects: All subjects enrolled into the study with intent to treat with the Axium Neurostimulator for the Management of Chronic Neuropathic Pain of the Foot and/or Lower Leg
Period: Overall Study
Arm/Group | All Enrolled Subjects
Started | 10
Received Trial System | 9
Receiving Permanent System | 8
Completed | 0
Not Completed | 10
Not completed — Sponsor terminated study | 4
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 2
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled Subjects: All subjects enrolled into the study with intent to treat with the Axium Neurostimulator
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 54 [25 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity for Overall Pain From Pre-treatment Baseline
Description: The Visual Analog Scale (VAS) is self-administered instrument assessing average pain intensity. Subjects rated their pain on a horizontal line, 10 cm in length, anchored by word descriptors on each end (no pain to worst imaginable pain). A higher score indicates a higher pain level. The values range from 0 (minimum) to 10 (maximum).
Time Frame: Baseline, 3, 6 and12-Months
Population: Differences in participants over time is due to early withdrawals and missing data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 8
units on a scale
  Baseline | 8.0 (1.5)
  3-Months: number analyzed (Participants) | 4
  3-Months | 4.7 (3.2)
  6-Months: number analyzed (Participants) | 4
  6-Months | 6.4 (2.3)
  12-Months: number analyzed (Participants) | 2
  12-Months | 5.4 (0.3)

ADVERSE EVENTS:
Time Frame: All adverse events reported spontaneously by the subject or observed by the investigator or his staff were recorded from the time of enrollment to study completion or early withdrawal.
Arm/Group | All Enrolled Subjects
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects (N=10)
Central disc hernia at L5-S1 and discreet bulging at L4-L5 (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects (N=10)
Headache and nausea (Injury, poisoning and procedural complications) | 1 (1) — These Adverse Events were monitored/assessed in such a manner that the specific Adverse Event Terms cannot be separated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days